CLINICAL TRIAL: NCT07406360
Title: A Phase 3a, Observer Blind, Randomized, Controlled Study to Evaluate the Immunogenicity and Safety of Intramuscular Administration of an Investigational Combined Measles, Mumps, Rubella, and Varicella Vaccine Compared With Intramuscular Administration of ProQuad When Administered as a Second Dose to Healthy Children Aged 15 Months to 6 Years of Age
Brief Title: A Study on the Immune Response and Safety of an Investigational Combined Measles, Mumps, Rubella and Varicella Vaccine, When Administered as Intramuscular Injection to Healthy Children 15 Months to 6 Years of Age
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 224349; 2025-523274-17-00 (Other: EU CT Number)
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Measles
Keywords: Measles; Mumps; Rubella; Varicella; Safety; Immunogenicity
MeSH Terms: conditions — Measles; Mumps; Rubella; Chickenpox | interventions — Chickenpox Vaccine; measles, mumps, rubella, varicella vaccine; Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study is observer-blind, participants care providers investigators and outcomes assessors are blinded but Investigational Medicinal Product administrators are unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MMRVNS Group (Experimental): Children, 15 months to 6 years old, who will receive one dose of MMRVNS on Day 1.
  Interventions: Biological: MMRVNS
- MMRV Group (Active Comparator): Children, 15 months to 6 years old, who will receive one dose of MMRV on Day 1.
  Interventions: Biological: MMRV

INTERVENTIONS:
Biological: MMRVNS — One dose of MMRVNS administered intramuscularly.
  Other Names: Investigational measles, mumps, rubella and varicella vaccine
  Arms: MMRVNS Group
Biological: MMRV — One dose of MMRV administered intramuscularly.
  Other Names: Merck's measles, mumps, rubella and varicella (ProQuad) vaccine
  Arms: MMRV Group

SUMMARY:
This study is evaluating the immunogenicity and safety of intramuscular administration of the investigational MMRVNS vaccine compared to intramuscular administration of the MMRV (Merck's measles, mumps, rubella and varicella) vaccine (ProQuad) that is already licensed for this route, when administered as a second dose in children 15 months to 6 years of age who were previously primed with a first dose of any combination of measles, mumps, rubella and varicella-containing vaccine(s).

ELIGIBILITY:
Inclusion Criteria:

* Participants' parent(s)/legally acceptable representative(s) (LAR(s)) who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written or witnessed/thumb printed informed consent obtained from the participants parent(s)/LAR(s) prior to performance of any study specific procedure.
* Informed assent obtained from the participants in line with local rules and regulations.
* Healthy participants as established by medical history and clinical examination at screening.

For countries where the second dose of measles, mumps, rubella, and varicella vaccination is administered between 4 and 6 years of age:

* A male or female participant between and including 4 and 6 years of age at the time of the study intervention administration, and in accordance with local regulations.
* Participant who previously received a first dose of varicella-containing vaccine in the second year of life.
* Participant who previously received a first dose of measles, mumps, rubella-containing vaccine in the second year of life.

For other countries:

* A male or female participant between and including 15 months to 6 years of age at the time of study intervention administration, and in accordance with local regulations.
* Participant who previously received a first dose of varicella-containing vaccine in the second year of life, or earlier at 11 months of age in accordance with national vaccination schedule following official recommendation, at least 3 months before study entry.
* Participant who previously received a first dose of measles, mumps, rubella-containing vaccine in the second year of life, or earlier at 11 months of age in accordance with national vaccination schedule following official recommendation, at least 1 month before study entry.

Exclusion Criteria:

Medical conditions

* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study interventions, including hypersensitivity to neomycin or, gelatin.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Hypersensitivity to latex.
* Unstable chronic conditions as determined by medical history and physical examination.
* Major congenital defects, as assessed by the investigator.
* History of measles, mumps, rubella, or varicella/zoster disease, as evaluated by the investigator.
* Recurrent history or uncontrolled neurological disorders or any neuroinflammatory, congenital neurological conditions, encephalopathies, or seizures.
* History of febrile seizures, for participant under 4 years of age.
* Active untreated tuberculosis.
* Condition that, in the judgement of the investigator, would make intramuscular injection unsafe.
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the clinical study.

Prior/Concomitant therapy

* Use of any investigational or non-registered product other than the study interventions during the period beginning 30 days before the dose of study intervention, or their planned use during the study period.
* Administration of immunoglobulins or other blood products or plasma derivates during the period starting 90 days before the study intervention or planned administration during the study period.
* Chronic administration of immune-modifying drugs (defined as more than 14 consecutive days in total) and/or planned use of long-acting immune-modifying treatments at any time up to the end of the study.

  * Up to 90 days prior to the study interventions administration: systemic corticosteroid.
  * Up to 180 days prior to study intervention administration: long-acting immune-modifying drugs including among others immunotherapy, monoclonal antibodies, antitumoral medication.
* Previous vaccination with a second dose of varicella containing vaccine or measles, mumps, rubella-containing vaccine.
* Use of salicylates or salicylate-containing products or its planned use during the period of 6 weeks following study intervention administration.
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the dose and ending 43 days after the dose of study intervention administration, with the exception of:
* Inactivated influenza vaccine, which may be given at any time during the study and administered at a different location than the study intervention, and
* Diphtheria, tetanus, acellular pertussis-containing vaccines may be administrated according to the local immunization practices of each participating country. It has to be administered on the same day as the study intervention administration at a different location. However, other than protocol-specified DTaP brand and diphtheria, tetanus, whole cell pertussis-containing vaccines are not allowed.

If emergency mass vaccination for an unforeseen public health threat is recommended and/or organized by public health authorities outside the routine immunization program, the time period described above can be reduced provided it is used according to the local governmental recommendations and sponsor is notified.

Prior/Concurrent clinical study participation

• Concurrently participating in another clinical study, at any time during the study period,

Other exclusion criteria

* Any study personnel's immediate dependents, family, or household members.
* Child in care.
* Participants with the following high-risk individuals in their household:

  * Immunocompromised individuals.
  * Pregnant women without documented history of varicella.
  * Newborn infants of mothers without documented history of varicella.
  * Newborn infants born <28 weeks of gestation.

Ages: 15 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1209 (Estimated)
Dates: Start 2026-04-13 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-06-22 (Estimated)

PRIMARY OUTCOMES:
Seroresponse of Immunoglobulin G (IgG) concentrations against measles | At Day 43
Seroresponse of IgG concentrations against mumps | At Day 43
Seroresponse of IgG concentrations against rubella | At Day 43
Seroresponse of IgG concentrations against Varicella zoster virus (VZV) | At Day 43
IgG concentrations against measles | At Day 43
IgG concentrations against mumps | At Day 43
IgG concentrations against rubella | At Day 43
IgG concentrations against VZV | At Day 43

SECONDARY OUTCOMES:
Number of participants with any solicited administration site events | From Day 1 to Day 4 for injection site redness, pain/tenderness and swelling; and from Day 1 to Day 43 for injection site varicella-like rash
  Solicited administration site events are injection site redness, pain/tenderness, swelling, and injection site varicella-like rash.
Number of participants with any solicited systemic events | From Day 1 to Day 15 for somnolence and loss of appetite; Day 1 to Day 22 for fever; and Day 1 to Day 43 for varicella-like rash, measles/rubella-like rash and other rash
  Solicited systemic events are somnolence (sleepiness/drowsiness), loss of appetite, fever, non-injection site varicella-like rash, measles/rubella-like rash and other rash.
Number of participants with any unsolicited adverse events (AEs) | From Day 1 up to Day 43 (during the 43 days following study intervention administration)
Number of participants with any medically attended adverse events (MAAEs) | From Day 1 up to Day 181 (during the 181 days following study intervention administration)
Number of participants with any serious AEs (SAEs), fatal SAEs, related SAEs | From Day 1 up to study end (Day 181)

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf